CLINICAL TRIAL: NCT01724034
Title: Daily Lung Ultrasound Assisting Weaning From Mechanical Ventilation in Difficult-to-wean Adult Patients - a Randomized Trial.
Brief Title: Lung Ultrasound Assisting Weaning in Difficult-to-wean Patients
Acronym: WeanUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Ernesto Dornelles (Other)
Collaborators: Hospital Moinhos de Vento (Other); Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Felippe Leopoldo Dexheimer Neto, M.D., Hospital Ernesto Dornelles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 094/2011
Record Dates: First submitted 2012-11-05; First posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Difficult-to-wean Adult Patients
Keywords: Weaning; Mechanical Ventilation; Lung Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily Lung Ultrasound (Experimental): If there is no lung sliding - evaluation for pneumothorax or mainstream intubation.
  If lung ultrasound shows normal pattern - search for reversible airway obstruction or venous embolism. If the patient has COPD, non invasive ventilation must be used as mode of discontinuing mechanical ventilation.
  If lung ultrasound shows intersticial syndrome - evaluate the need to negativate hydric balance before the next spontaneous breathing trial.
  If findings are asymmetrical - search for new or uncontrolled infection. If there is simple pleural effusion - researchers should determine a negativation of hydric balance or perform thoracocentesis.
  If there are signs of complicated pleural effusion - a new image technique should be performed as evaluated by the surgical team.
  Interventions: Other: Abolish Lung Sliding; Other: Normal Lung Ultrasound; Other: Pulmonary Interstitial Syndrome; Other: Asymmetrical Lung Ultrasound; Other: Simple Pleural Effusion; Other: Complex Pleural Effusion
- Control Group (No Intervention)

INTERVENTIONS:
Other: Abolish Lung Sliding — If there is no lung sliding, the patient will be promptly evaluated for pneumothorax or mainstream intubation.
  Arms: Daily Lung Ultrasound
Other: Normal Lung Ultrasound — If the patient fails the spontaneous breathing trial and the lung ultrasound examination is normal - researchers will investigate venous thrombosis (deep vein thrombosis and/or pulmonary embolism) and rule out reversible airway obstruction. If the patient has the previous diagnosis of COPD, non invasive mechanical ventilation is indicated for facilitate weaning.
  Arms: Daily Lung Ultrasound
Other: Pulmonary Interstitial Syndrome — If lung ultrasound shows "B pattern" - cardiogenic pulmonary edema will be differentiated from Acute Respiratory Distress Syndrome (ARDS). If cardiogenic edema is a possibility, diuretics will be administrated (at least 40 mg of furosemide) or ultrafiltration will be performed. The main target is a negative fluid balance of, at least, 1000 ml before the next spontaneous breathing trial. Another possibility is to titrate vasodilators (at least a 20% reduction in the systolic blood pressure) before the next spontaneous breathing trial.
  Other Names: B Lines
  Arms: Daily Lung Ultrasound
Other: Asymmetrical Lung Ultrasound — If lung ultrasound shows asymmetrical findings, the occurence of new or uncontrolled infection (pulmonary or extrapulmonary) will be investigated.
  Other Names: AB Profile or Consolidation
  Arms: Daily Lung Ultrasound
Other: Simple Pleural Effusion — If the patient has pleural effusion without ultrasonographic signs of complications (any hyperechoic pattern or complex septated pattern), researchers will administrate diuretics (at least 40 mg of furosemide in 24 hours) or increase ultrafiltration - to achieve a negative fluid balance of, at least, 1000 ml before the next spontaneous breathing trial. Another possibility is to perform pleural drainage.
  Arms: Daily Lung Ultrasound
Other: Complex Pleural Effusion — If there is pleural effusion with hyperechoic or septated pattern, another image exam will be performed and evaluated by the surgical team.
  Arms: Daily Lung Ultrasound

SUMMARY:
Daily lung ultrasound can help weaning from mechanical ventilation in difficult-to-wean adult patients. In this randomized trial, standardized lung ultrasound will be performed daily asssociated with standardized interventions aiming to decrease the total time in mechanical ventilation.

DETAILED DESCRIPTION:
This trial will be performed in two intensive care units (ICUs). After randomization, all patients in the intervention group will undergo daily lung ultrasounds before the next spontaneous breathing trial. The results from the lung ultrasound will indicate specific interventions to facilitate weaning:

* No sign of lung sliding (ultrasound finding suggestive of pleural movement): prompt evaluation for pneumothorax or mainstream intubation will be indicated;
* normal lung ultrasound (ultrasound A profile): the patient will be evaluated for deep vein thrombosis / pulmonary embolism and/or for reversible airway obstruction (e.g. uncontrolled asthma or COPD [Chronic Obstructive Pulmonary Disease] exacerbation)- followed by appropriate treatment. If the patient has COPD, non invasive mechanical ventilation must be used as mode of discontinuing mechanical ventilation;
* lung ultrasound shows pulmonary edema (ultrasound B profile): cardiogenic pulmonary edema will be differentiated from acute Respiratory Distress Syndrome (ARDS) - followed by appropriate treatment (e.g. a negative fluid balance of, at least, 1000 ml before the next spontaneous breathing trial);
* lung ultrasound shows asymmetrical patterns (ultrasound AB profile or Pulmonary Consolidation): the possibility of an uncontrolled infection will be investigated;
* presence of simple pleural effusion: diuretics will be indicated (for a negative fluid balance of, at least, 1000 ml before the next spontaneous breathing trial) or thoracocentesis at description of the assistant team;
* presence of complex pleural effusion: other image exam will be performed, and will be evaluated by the surgical team.

ELIGIBILITY:
Inclusion Criteria:

* Difficult to Wean;
* 1 failure in the spontaneous breathing trial or 1 extubation failure
* Adult patients (over 18 years old);

Exclusion Criteria:

* Palliative Care;
* Life expectancy under 90 days;
* COPD Gold IV, Cirrhosis Child C, Metastatic Cancer with low performance, etc
* Other weaning method than institutional protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Time in mechanical ventilation | from intubation until extubation success (defined as weaning from mechanical support for, at least, 48 hours) or death (days)

SECONDARY OUTCOMES:
Number of tracheostomies performed | patients follow-up will continue until weaning from mechanical support, up to 2 months
Length of ICU stay | from icu admition until icu discharge, up to 2 months
Incidence of ventilation-associated pneumonia | until icu discharge, up to 2 months
ICU's, Hospital's and 28-days mortality | until ICU's and hospital's discharge and 28th day from ICU admisson, with an expected average of 4 weeks
Performance status at ICU's and Hospital's discharge | at icu's and hospital discharge, with an expected average of 4 weeks
Correlation between findings from ultrasound and other image techniques | after data collection (1 year) - retrospective review
Duration of Weaning | From first failed spontaneous breathing trial or failed extubation until weaning from mechanical ventilation support, up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Felippe L Dexheimer, MD, Principal Investigator — Hospital Ernesto Dornelles; Cassiano Teixeira, MD, PhD, Study Chair — Hospital Moinhos de Vento; Paulo R Dalcin, MD, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul, Brazil